CLINICAL TRIAL: NCT07381270
Title: Simulation-Based Team Training to Improve Psychological Safety and Relational Coordination in Clinical Teams
Brief Title: Using Simulation-based Team Training to Improve Psychological Safety and Relational Coordination as Well as Conducting a Process Evaluation
Acronym: InfecSIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: InfecSIM
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-03

CONDITIONS: Medical Education, Simulation, Crisis Resource Management; Simulation Training; Simulation Based Medical Education; Culture
Keywords: Simulation-based team training; relational coordination; psychologically safety

STUDY DESIGN:
Intervention Model Description: A controlled intervention study comparing two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation intervention (Experimental)
  Interventions: Behavioral: Simulation-based team training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Simulation-based team training — Staff participates in a simulation-based training initiative
  Arms: Simulation intervention

SUMMARY:
Simulation-based team training is increasingly used in hospitals to support teamwork and communication, particularly in situations that are complex or time-critical. While such training is known to improve observable team behaviours, less is known about how it is implemented in everyday clinical work and how it influences relational aspects of teamwork, such as psychological safety and relational coordination.

This study explores the implementation and perceived impact of a simulation-based training programme focused on infectious disease management in a hospital department. Psychological safety refers to whether staff feel safe to speak up, ask questions, and express concerns, while relational coordination concerns how well different professional groups communicate, share goals, and align their work.

Using a qualitative process and outcome evaluation, the study examines how the simulation activities were introduced, adapted, and experienced by different staff groups, and how participants perceived their influence on collaboration and professional behaviour. Data are collected through interviews with clinical staff and managers, questionnaires measuring psychological safety and relational coordination before and after the intervention, and systematic registration of simulation activities (including who participated, what was trained, and when and where simulations took place).

By combining process evaluation with an exploration of perceived outcomes, the study aims to provide insight into how simulation-based team training functions as a behavioural intervention in complex clinical settings, and how it may support psychologically safe and well-coordinated teamwork in everyday practice.

ELIGIBILITY:
Inclusion Criteria:

* Employed in the included departments
* Profession as a doctor or nurse

Exclusion Criteria:

* If participants are employed in both intervention and control group during the project period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Psychological safety | Baseline and immediately after the intervention period.
  Psychological safety will be assessed using the Team Psychological Safety scale (Edmondson). The scale consists of 7 items rated on a 1-7 Likert scale, with higher scores indicating greater psychological safety. The outcome will be reported as the mean questionnaire score. Qualitative interviews are not included in this outcome measure.
Relational coordination | Baseline and immediately after the intervention period.
  Relational coordination will be assessed using the Relational Coordination Survey (Gittell). Items are rated on a 1-5 scale, with higher scores indicating stronger relational coordination. The outcome will be reported as the mean questionnaire score. Qualitative interviews are not included in this outcome measure.

OTHER OUTCOMES:
Process evaluation | From intervention start until immediately after the intervention period.
  The process evaluation examines how the simulation-based team training was implemented, including organisation, adaptation, and contextual conditions shaping delivery and participation. Data are collected through qualitative interviews and systematic registration of simulation activities.
Qualitative explanatory evaluation of intervention mechanisms | Immediately after the intervention period.
  Qualitative interviews will explore how staff and managers describe changes in everyday work practices following the simulation-based team training and how these changes are understood within the local clinical context. Outcomes will be reported as qualitative themes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No